CLINICAL TRIAL: NCT01462357
Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' HPV-16/18 L1 AS04 Vaccine and Merck's Gardasil Vaccine When Administered According to Alternative 2-dose Schedules in 9-14 Year Old Females
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' Human Papillomavirus (HPV) Vaccine (GSK-580299) and Merck's Gardasil Vaccine When Administered According to Alternative 2-dose Schedules in 9-14 Year Old Females
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 115411; 2011-002035-26 (EudraCT Number)
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Infections, Papillomavirus
Keywords: Human papillomavirus; Safety; HPV vaccine; Immune response
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Cervarix 2 dose Group (Experimental): Subjects who received 2 doses of Cervarix vaccine at Day 0 and Month 6 and 1 dose of placebo at Month 2. The vaccines were administered intramuscularly, in the deltoid muscle of the non-dominant upper arm.
  Interventions: Biological: Cervarix; Drug: Placebo
- Gardasil 2 dose Group (Experimental): Subjects who received 2 doses of Gardasil vaccine at Day 0 and Month 6 and 1 dose of placebo at Month 2. The vaccines were administered intramuscularly, in the deltoid muscle of the non-dominant upper arm.
  Interventions: Biological: Gardasil; Drug: Placebo
- Gardasil 3 dose Group (Experimental): Subjects who received 3 doses of Gardasil vaccine at Day 0 and at Months 2 and 6. The vaccines were administered intramuscularly, in the deltoid muscle of the non-dominant upper arm.
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: Cervarix — 2 doses of 0.5 mL supplied as a liquid in individual pre-filled syringes to be administered intramuscularly in the deltoid muscle of the non-dominant arm at Day 0 and Month 6.
  Arms: Cervarix 2 dose Group
Biological: Gardasil — 2 or 3 doses of 0.5 mL supplied as a liquid in individual pre-filled syringes or vials to be administered intramuscularly in the deltoid muscle of the non-dominant arm at Day 0 and Month 6 (Gardasil 2 dose Group) or at Day 0, Month 2 and Month 6 (Gardasil 3 dose Group), respectively.
  Arms: Gardasil 2 dose Group; Gardasil 3 dose Group
Drug: Placebo — 2 doses of 0.5 mL supplied as a liquid in individual pre-filled syringes to be administered intramuscularly in the deltoid muscle of the non-dominant arm at Month 2 to maintain blinding.
  Arms: Cervarix 2 dose Group; Gardasil 2 dose Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and the safety of Cervarix administered according to a 2-dose schedule at 0, 6 months compared to Gardasil, administered according to a 2-dose schedule at 0, 6 months or the standard 3-dose schedule of 0, 2, 6 months in 9-14 years old healthy females.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol and subjects who the investigator believes their parent(s)/Legally Acceptable Representative(s) (LAR[s]) can and will comply with the requirements of the protocol.
* A female between, and including, 9 and 14 years of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to enrolment in the study. In addition, if capable, the subject should sign and personally date a written informed assent.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for two months after completion of the vaccination series.

Exclusion Criteria:

* Pregnant or breastfeeding.
* A woman planning to become pregnant, likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the vaccination phase of the study, i.e. up to two months after the last vaccine dose.
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study other than those foreseen in the protocol.
* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period (up to Month 36).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccines.
* Cancer or autoimmune disease under treatment.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before each dose of vaccine. Administration of routine meningococcal, hepatitis B, hepatitis A, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before each dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous administration of vaccine components.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests, which in the opinion of the investigator precludes administration of the study vaccine.
* Acute disease and/or fever at the time of enrolment.
* Drug and/or alcohol abuse.

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1079 (Actual)
Dates: Start 2011-11-21 (Actual); Primary Completion 2015-10-27 (Actual); Study Completion 2015-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- France (10):
  - GSK Investigational Site, Dax
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Saint Cyr Sur Loir
  - GSK Investigational Site, Seysses
  - GSK Investigational Site, Tours
- Hong Kong (2):
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- GSK Investigational Site, Singapore, Singapore
- Sweden (3):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Örebro

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below).
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=4513

REFERENCES:
- [Background] Leung TF, Liu AP, Lim FS, Thollot F, Oh HM, Lee BW, Rombo L, Tan NC, Rouzier R, Friel D, De Muynck B, De Simoni S, Suryakiran P, Hezareh M, Folschweiller N, Thomas F, Struyf F. Comparative immunogenicity and safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine and HPV-6/11/16/18 vaccine administered according to 2- and 3-dose schedules in girls aged 9-14 years: Results to month 12 from a randomized trial. Hum Vaccin Immunother. 2015;11(7):1689-702. doi: 10.1080/21645515.2015.1050570. PMID 26062002
- [Background] Leung TF, Liu AP, Lim FS, Thollot F, Oh HML, Lee BW, Rombo L, Tan NC, Rouzier R, De Simoni S, Suryakiran P, Hezareh M, Thomas F, Folschweiller N, Struyf F. Comparative immunogenicity and safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine and 4vHPV vaccine administered according to two- or three-dose schedules in girls aged 9-14 years: Results to month 36 from a randomized trial. Vaccine. 2018 Jan 2;36(1):98-106. doi: 10.1016/j.vaccine.2017.11.034. Epub 2017 Nov 23. PMID 29174109
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 115411 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115411 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115411 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115411 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115411 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115411 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1079 subjects entered this study, of which 4 subjects signed an informed consent but did not receive a single dose of the vaccine and were hence not counted as starting the study.
Period: Overall Study
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Started | 359 | 358 | 358
Completed | 351 | 339 | 346
Not Completed | 8 | 19 | 12
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 11 | 3
Not completed — Migrated/moved from study area | 2 | 3 | 1
Not completed — Lost to Follow-up | 3 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group | Total
Number analyzed (Participants) | 359 | 358 | 358 | 1075
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.5 (1.64) | 11.5 (1.56) | 11.6 (1.64) | 11.53 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 359 | 358 | 358 | 1075
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 4 | 6 | 4 | 14
  Asian - Central / South Asian Heritage | 1 | 1 | 2 | 4
  Asian - East Asian Heritage | 179 | 178 | 179 | 536
  Asian - South East Asian Heritage | 81 | 78 | 83 | 242
  White - Arabic / North African Heritage | 5 | 7 | 7 | 19
  White - Caucasian / European Heritage | 89 | 86 | 83 | 258
  White - Caucasian / African Heritage | 0 | 1 | 0 | 1
  African - White / Caucasian Heritage | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Anti-HPV-16/18 Antibodies as Assessed by Enzyme-Linked Immunosorbent Assay (ELISA) at Month 7 Based on the ATP Cohort for Immunogenicity
Description: Seroconversion was defined as the appearance of antibodies (i.e. anti-HPV-16 and anti-HPV-18 antibody titers greater than or equal to (≥) 19 and 18 ELISA units per milliliter (EL.U/mL), respectively), in the serum of subjects seronegative before vaccination.
Time Frame: At Month 7 (i.e. one month after the last dose of study vaccine)
Population: The analysis was based on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available at the specified time point and who were seronegative before vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 334 | 331 | 333
Participants
  Anti-HPV-16: number analyzed (Participants) | 330 | 327 | 322
  Anti-HPV-16 | 330 | 327 | 322
  Anti-HPV-18 | 334 | 331 | 333
Statistical Analysis 1: Comparison: Cervarix 2 Dose Group vs Gardasil 2 Dose Group; Immune response to anti-HPV-16 in terms of seroconversion rates (SCR): To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule at 0, 6 months is non-inferior to that of Gardasil vaccine administered according to a 2-dose schedule at 0, 6 months, 1 month after the last dose (Month 7), in initially seronegative subjects; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion was shown if, one month after the last dose, for both anti-HPV-16 and anti-HPV-18 antibodies, the upper limit of the 95% confidence interval (CI) for the difference (Gardasil 2 dose Group minus Cervarix 2 dose Group) was below 5%; Difference in SCR = 0, 95% CI 2-sided [-1.16 to 1.15]
Statistical Analysis 2: Comparison: Cervarix 2 Dose Group vs Gardasil 2 Dose Group; Immune response to anti-HPV-18 in terms of SCR: To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule at 0, 6 months is non-inferior to that of Gardasil vaccine administered according to a 2-dose schedule at 0, 6 months, 1 month after the last dose (Month 7), in initially seronegative subjects; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in SCR = 0, 95% CI 2-sided [-1.15 to 1.14]

2. Primary Outcome: Anti-HPV-16/18 Antibody Titers as Assessed by ELISA at Month 7 Based on the ATP Cohort for Immunogenicity
Description: Anti-HPV 16/18 antibody titers were presented as Geometric Mean Titers (GMTs) and expressed in EL.U/mL.
Time Frame: At Month 7 (i.e. one month after the last dose of study vaccine)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 334 | 331 | 333
EL.U/mL
  Anti-HPV-16: number analyzed (Participants) | 330 | 327 | 322
  Anti-HPV-16 | 8244.1 [7678.3 to 8851.7] | 5056.0 [4596.5 to 5561.5] | 4807.4 [4420.8 to 5227.7]
  Anti-HPV-18 | 5277.4 [4858.6 to 5732.4] | 1207.2 [1092.9 to 1333.4] | 1653.5 [1484.4 to 1841.8]
Statistical Analysis 1: Comparison: Cervarix 2 Dose Group vs Gardasil 2 Dose Group; Immune response to anti-HPV-16 in terms of Geometric Mean Titers (GMT): To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule at 0, 6 months is non-inferior to that of Gardasil vaccine administered according to a 2-dose schedule at 0, 6 months, 1 month after the last dose (Month 7), in initially seronegative subjects; Test type: Non-Inferiority — Non-inferiority with respect to GMT was shown if, one month after the last dose, for both anti-HPV-16 and anti-HPV-18 antibodies, the upper limit of the 95% CI for the GMT ratio (Gardasil 2 dose Group divided by Cervarix 2 dose Group) was below 2; ANOVA; GMT ratio = 0.61, 95% CI 2-sided [0.54 to 0.69]
Statistical Analysis 2: Comparison: Cervarix 2 Dose Group vs Gardasil 2 Dose Group; Immune response to anti-HPV-18 in terms of GMT: To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule at 0, 6 months is non-inferior to that of Gardasil vaccine administered according to a 2-dose schedule at 0, 6 months, 1 month after the last dose (Month 7), in initially seronegative subjects; Test type: Non-Inferiority — Non-inferiority with respect to GMT was shown if, one month after the last dose, for both anti-HPV-16 and anti-HPV-18 antibodies, the upper limit of the 95% confidence interval (CI) for the GMT ratio (Gardasil 2 dose Group divided by Cervarix 2 dose Group) was below 2; ANOVA; GMT ratio = 0.23, 95% CI 2-sided [0.20 to 0.26]

3. Primary Outcome: Anti-HPV-16/18 Antibody Titers as Assessed by ELISA at Month 7 Based on the Total Vaccinated Cohort (TVC)
Description: Anti-HPV 16/18 antibody titers were presented as Geometric Mean Titers (GMTs) and expressed in EL.U/mL.
Time Frame: At Month 7 (i.e. one month after the last dose of study vaccine)
Population: The analysis was based on the TVC which included all subjects, regardless of serostatus, who received at least one dose of vaccine in this study and for whom data were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 357 | 353 | 351
EL.U/mL
  Anti-HPV-16 | 8256.4 [7650.3 to 8910.6] | 4886.1 [4435.4 to 5382.6] | 4789.2 [4409.6 to 5201.4]
  Anti-HPV-18 | 5267.8 [4857.1 to 5713.2] | 1166.3 [1056 to 1288.2] | 1635.8 [1470 to 1820.4]
Statistical Analysis 1: Comparison: Cervarix 2 Dose Group vs Gardasil 2 Dose Group; Anti-HPV-18 immune response: To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule at 0, 6 months is superior to that of Gardasil vaccine administered according to a 2-dose schedule at 0, 6 months, in 9-14 year-old females, 1 month after the last dose (Month 7) regardless of serostatus; Test type: Superiority — Superiority was shown if the lower limit of the 95% CI for the ratio of GMTs (Cervarix 2 dose Group divided by Gardasil 2 dose Group) was above 1 for anti-HPV-18 antibodies; p = 0.0001, ANOVA; GMT ratio = 4.52, 95% CI 2-sided [3.97 to 5.13]
Statistical Analysis 2: Comparison: Cervarix 2 Dose Group vs Gardasil 2 Dose Group; Anti-HPV-16 immune response: To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule at 0, 6 months is superior to that of Gardasil vaccine administered according to a 2-dose schedule at 0, 6 months, in 9-14 year-old females, 1 month after the last dose (Month 7) regardless of serostatus; Test type: Superiority — Superiority was shown if the lower limit of the 95% CI for the ratio of GMTs (Cervarix 2 dose Group divided by Gardasil 2 dose Group) was above 1 for anti-HPV-16 antibodies; p = 0.0001, ANOVA; GMT ratio = 1.69, 95% CI 2-sided [1.49 to 1.91]

4. Secondary Outcome: Anti-HPV-16/18 Seroconversion Rates as Assessed by ELISA
Description: Seroconversion was defined as the appearance of antibodies (i.e. anti-HPV-16 and anti-HPV-18 antibody titers ≥ 19 and 18 EL.U/mL, respectively) in the serum of subjects seronegative before vaccination.
Time Frame: At Day 0 and Months 12, 18, 24 and 36
Population: The analysis was based on the Month 36 ATP cohort for immunogenicity, which included subjects who returned for blood sampling at Month 36, for whom data concerning immunogenicity outcome measures were available at the specified time points and who were seronegative before vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 322 | 310 | 320
Participants
  Anti-HPV-16, Day 0: number analyzed (Participants) | 318 | 306 | 309
  Anti-HPV-16, Day 0 | 0 | 0 | 0
  Anti-HPV-18, Day 0 | 0 | 0 | 0
  Anti-HPV-16, Month 12: number analyzed (Participants) | 317 | 305 | 308
  Anti-HPV-16, Month 12 | 316 | 305 | 308
  Anti-HPV-18, Month 12: number analyzed (Participants) | 321 | 309 | 319
  Anti-HPV-18, Month 12 | 320 | 309 | 319
  Anti-HPV-16, Month 18: number analyzed (Participants) | 316 | 305 | 309
  Anti-HPV-16, Month 18 | 316 | 304 | 309
  Anti-HPV-18, Month 18: number analyzed (Participants) | 320 | 309 | 320
  Anti-HPV-18, Month 18 | 320 | 294 | 313
  Anti-HPV-16, Month 24: number analyzed (Participants) | 314 | 304 | 307
  Anti-HPV-16, Month 24 | 314 | 303 | 307
  Anti-HPV-18, Month 24: number analyzed (Participants) | 318 | 308 | 318
  Anti-HPV-18, Month 24 | 318 | 287 | 308
  Anti-HPV-16, Month 36: number analyzed (Participants) | 318 | 306 | 309
  Anti-HPV-16, Month 36 | 318 | 304 | 308
  Anti-HPV-18, Month 36 | 322 | 267 | 297

5. Secondary Outcome: Anti-HPV-16/18 Antibody Titers as Assessed by ELISA
Description: Anti-HPV 16/18 antibody titers were presented as GMTs and expressed in EL.U/mL based on ELISA.
Time Frame: At Day 0 and Months 12, 18, 24 and 36
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 322 | 310 | 320
EL.U/mL
  Anti-HPV-16, Day 0: number analyzed (Participants) | 318 | 306 | 309
  Anti-HPV-16, Day 0 | 9.5 [9.5 to 9.5] | 9.5 [9.5 to 9.5] | 9.5 [9.5 to 9.5]
  Anti-HPV-18, Day 0 | 9.0 [9.0 to 9.0] | 9.0 [9.0 to 9.0] | 9.0 [9.0 to 9.0]
  Anti-HPV-16, Month 12: number analyzed (Participants) | 317 | 305 | 308
  Anti-HPV-16, Month 12 | 2209.2 [2014 to 2423.4] | 1294.8 [1160.4 to 1444.9] | 1600.7 [1457.3 to 1758.2]
  Anti-HPV-18, Month 12: number analyzed (Participants) | 321 | 309 | 319
  Anti-HPV-18, Month 12 | 1299.3 [1176.2 to 1435.6] | 266.6 [236.3 to 300.8] | 478.5 [422.8 to 541.6]
  Anti-HPV-16, Month 18: number analyzed (Participants) | 316 | 305 | 309
  Anti-HPV-16, Month 18 | 1488.8 [1365.5 to 1623.3] | 684.4 [605.8 to 773.2] | 824.0 [744.4 to 912.2]
  Anti-HPV-18, Month 18: number analyzed (Participants) | 320 | 309 | 320
  Anti-HPV-18, Month 18 | 754.2 [682.6 to 833.2] | 134.8 [118.1 to 154] | 231.3 [202.4 to 264.4]
  Anti-HPV-16, Month 24: number analyzed (Participants) | 314 | 304 | 307
  Anti-HPV-16, Month 24 | 1285.0 [1181.1 to 1398.0] | 514.1 [455.4 to 580.3] | 637.1 [575.8 to 704.9]
  Anti-HPV-18, Month 24: number analyzed (Participants) | 318 | 308 | 318
  Anti-HPV-18, Month 24 | 613.7 [555.0 to 678.6] | 106.3 [93.2 to 121.3] | 182.0 [159.3 to 208.0]
  Anti-HPV-16, Month 36: number analyzed (Participants) | 318 | 306 | 309
  Anti-HPV-16, Month 36 | 1061.4 [971.8 to 1159.4] | 379.8 [333.4 to 432.7] | 472.4 [425 to 525.0]
  Anti-HPV-18, Month 36 | 486.5 [437.8 to 540.6] | 71.0 [62.0 to 81.2] | 119.1 [103.4 to 137.1]

6. Secondary Outcome: Anti-HPV-16/18 Antibody Titers as Assessed by ELISA at Month 36
Description: Data at Month 36 were also expressed as International Units per milliliter (IU/mL). Conversion factor from EU/mL to IU/mL was determined to be 1/6.1 for HPV-16 and 1/5.7 for HPV-18, using the WHO International Standards (NIBSC codes 05-134 and 10-140 for HPV-16 and HPV-18, respectively). The assay cut-offs were therefore 3.1 IU/mL and 3.2 IU/mL for anti-HPV-16 and anti-HPV-18 antibodies, respectively.
Time Frame: At Month 36
Population: The analysis was based on the Month 36 ATP cohort for immunogenicity, which included subjects who returned for blood sampling at Month 36, for whom data concerning immunogenicity outcome measures were available at the specified time point and who were seronegative before vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 322 | 310 | 320
IU/mL
  Anti-HPV-16: number analyzed (Participants) | 318 | 306 | 309
  Anti-HPV-16 | 174.0 [159.3 to 190.1] | 62.3 [54.7 to 71.0] | 77.4 [69.6 to 86.0]
  Anti-HPV-18 | 85.3 [76.7 to 94.8] | 12.5 [10.9 to 14.3] | 20.9 [18.2 to 24.1]

7. Secondary Outcome: Anti-HPV-16/18 Seroconversion Rates as Assessed by Pseudovirion-based Neutralization Assay (PBNA) in a Subset of Subjects, Based on the Month 36 ATP Cohort for Immunogenicity
Description: Seroconversion was defined as the appearance of antibodies (i.e. anti-HPV-16 and anti-HPV-18 antibody titers ≥40 ED50) in the serum of subjects seronegative before vaccination. The assay was performed on a subset of approximately 100 subjects per study group.
Time Frame: At Day 0 and Months 7, 12, 18, 24 and 36
Population: The analysis was based on the Month 36 ATP cohort for immunogenicity, which included a subset of approximately 100 subjects per study group, who returned for blood sampling at Month 36, for whom immunogenicity data were available at the specified time point and who were seronegative before vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 89 | 87 | 91
Participants
  Anti-HPV-16, Day 0: number analyzed (Participants) | 89 | 85 | 91
  Anti-HPV-16, Day 0 | 0 | 0 | 0
  Anti-HPV-18, Day 0 | 0 | 0 | 0
  Anti-HPV-16, Month 7: number analyzed (Participants) | 89 | 85 | 91
  Anti-HPV-16, Month 7 | 89 | 85 | 91
  Anti-HPV-18, Month 7 | 89 | 87 | 91
  Anti-HPV-16, Month 12: number analyzed (Participants) | 88 | 85 | 91
  Anti-HPV-16, Month 12 | 88 | 85 | 91
  Anti-HPV-18, Month 12: number analyzed (Participants) | 88 | 87 | 91
  Anti-HPV-18, Month 12 | 88 | 86 | 91
  Anti-HPV-16, Month 18: number analyzed (Participants) | 88 | 85 | 90
  Anti-HPV-16, Month 18 | 88 | 83 | 89
  Anti-HPV-18, Month 18: number analyzed (Participants) | 87 | 87 | 91
  Anti-HPV-18, Month 18 | 87 | 77 | 89
  Anti-HPV-16, Month 24: number analyzed (Participants) | 86 | 83 | 91
  Anti-HPV-16, Month 24 | 86 | 83 | 90
  Anti-HPV-18, Month 24: number analyzed (Participants) | 86 | 83 | 91
  Anti-HPV-18, Month 24 | 86 | 75 | 88
  Anti-HPV-16, Month 36: number analyzed (Participants) | 89 | 85 | 91
  Anti-HPV-16, Month 36 | 89 | 85 | 91
  Anti-HPV-18, Month 36 | 89 | 75 | 86

8. Secondary Outcome: Anti-HPV-16/18 Antibody Titers as Assessed by PBNA in a Subset of Subjects, Based on the Month 36 ATP Cohort for Immunogenicity
Description: Anti-HPV 16/18 antibody titers were presented as GMT and expressed in titers using the PBNA. The assay was performed on a subset of approximately 100 subjects per study group.
Time Frame: At Day 0 and Months 7, 12, 18, 24 and 36
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 89 | 87 | 91
Titers
  Anti-HPV-16, Day 0: number analyzed (Participants) | 89 | 85 | 91
  Anti-HPV-16, Day 0 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Anti-HPV-18, Day 0 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Anti-HPV-16, Month 7: number analyzed (Participants) | 89 | 85 | 91
  Anti-HPV-16, Month 7 | 52868.5 [44171.0 to 63278.5] | 19130.1 [15166.8 to 24129.0] | 22182.7 [17611.7 to 27940.1]
  Anti-HPV-18, Month 7 | 24068.5 [19293.2 to 30025.8] | 4726.5 [3600.9 to 6204.0] | 8243.9 [6276.2 to 10828.4]
  Anti-HPV-16, Month 12: number analyzed (Participants) | 88 | 85 | 91
  Anti-HPV-16, Month 12 | 10695.9 [8564.9 to 13357.1] | 4280.1 [3245.9 to 5643.6] | 5843.8 [4599.8 to 7424.1]
  Anti-HPV-18, Month 12: number analyzed (Participants) | 88 | 87 | 91
  Anti-HPV-18, Month 12 | 3683.3 [2914.4 to 4655.2] | 689.0 [517.2 to 917.8] | 1788.6 [1308.6 to 2444.7]
  Anti-HPV-16, Month 18: number analyzed (Participants) | 88 | 85 | 90
  Anti-HPV-16, Month 18 | 8436.3 [6650.6 to 10701.4] | 2129.7 [1512.8 to 2998.1] | 2987.2 [2218.5 to 4022.3]
  Anti-HPV-18, Month 18: number analyzed (Participants) | 87 | 87 | 91
  Anti-HPV-18, Month 18 | 2426.3 [1885.7 to 3121.7] | 295.7 [217.0 to 402.8] | 812.1 [577.0 to 1143.0]
  Anti-HPV-16, Month 24: number analyzed (Participants) | 86 | 83 | 91
  Anti-HPV-16, Month 24 | 5036.7 [4097.8 to 6190.7] | 1211.8 [893.8 to 1642.9] | 1967.2 [1507.5 to 2567.2]
  Anti-HPV-18, Month 24: number analyzed (Participants) | 86 | 83 | 91
  Anti-HPV-18, Month 24 | 1763.0 [1384.5 to 2245.0] | 237.1 [177.2 to 317.1] | 573.1 [421.5 to 779.3]
  Anti-HPV-16, Month 36: number analyzed (Participants) | 89 | 85 | 91
  Anti-HPV-16, Month 36 | 4357.8 [3577.8 to 5307.9] | 1128.9 [857.4 to 1486.4] | 1577.0 [1210.4 to 2054.5]
  Anti-HPV-18, Month 36 | 1613.9 [1267.6 to 2054.7] | 185.8 [140.4 to 245.8] | 472.8 [345.8 to 646.4]

9. Secondary Outcome: Anti-HPV-16/18 Seroconversion Rates as Assessed by PBNA in a Subset of Subjects, Based on the Month 36 TVC
Description: as for outcome 7
Time Frame: At Day 0 and Months 7, 12, 18, 24 and 36
Population: The analysis was based on the Month 36 TVC, which included a subset of approximately 100 subjects per study group, who received at least one dose of vaccine in this study, for whom data were available at the specified time points and who were seronegative before vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 99 | 92 | 98
Participants
  Anti-HPV-16, Day 0: number analyzed (Participants) | 99 | 90 | 98
  Anti-HPV-16, Day 0 | 0 | 0 | 0
  Anti-HPV-18, Day 0 | 0 | 0 | 0
  Anti-HPV-16, Month 7: number analyzed (Participants) | 99 | 90 | 98
  Anti-HPV-16, Month 7 | 99 | 90 | 98
  Anti-HPV-18, Month 7 | 99 | 92 | 98
  Anti-HPV-16, Month 12: number analyzed (Participants) | 98 | 90 | 98
  Anti-HPV-16, Month 12 | 97 | 90 | 98
  Anti-HPV-18, Month 12: number analyzed (Participants) | 98 | 92 | 98
  Anti-HPV-18, Month 12 | 98 | 91 | 98
  Anti-HPV-16, Month 18: number analyzed (Participants) | 98 | 90 | 97
  Anti-HPV-16, Month 18 | 97 | 88 | 96
  Anti-HPV-18, Month 18: number analyzed (Participants) | 97 | 92 | 98
  Anti-HPV-18, Month 18 | 97 | 82 | 96
  Anti-HPV-16, Month 24: number analyzed (Participants) | 96 | 87 | 98
  Anti-HPV-16, Month 24 | 95 | 87 | 97
  Anti-HPV-18, Month 24: number analyzed (Participants) | 96 | 87 | 98
  Anti-HPV-18, Month 24 | 96 | 79 | 94
  Anti-HPV-16, Month 36: number analyzed (Participants) | 98 | 90 | 98
  Anti-HPV-16, Month 36 | 97 | 90 | 98
  Anti-HPV-18, Month 36: number analyzed (Participants) | 97 | 92 | 98
  Anti-HPV-18, Month 36 | 97 | 80 | 92

10. Secondary Outcome: Anti-HPV-16/18 Antibody Titers as Assessed by PBNA in a Subset of Subjects, Based on the Month 36 TVC
Description: as for outcome 8
Time Frame: At Day 0 and Months 7, 12, 18, 24 and 36
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 99 | 92 | 98
Titers
  Anti-HPV-16, Day 0: number analyzed (Participants) | 99 | 90 | 98
  Anti-HPV-16, Day 0 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Anti-HPV-18, Day 0 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Anti-HPV-16, Month 7: number analyzed (Participants) | 99 | 90 | 98
  Anti-HPV-16, Month 7 | 50000.7 [39742.9 to 62906.0] | 18573.7 [14876.8 to 23189.3] | 22294.2 [17763.8 to 27980.0]
  Anti-HPV-18, Month 7 | 23576.9 [18922.5 to 29376.2] | 4563.7 [3519.5 to 5917.8] | 8042.1 [6186.1 to 10454.8]
  Anti-HPV-16, Month 12: number analyzed (Participants) | 98 | 90 | 98
  Anti-HPV-16, Month 12 | 10039.6 [7884.1 to 12784.5] | 4174.9 [3207.5 to 5434.2] | 5766.0 [4573.8 to 7268.9]
  Anti-HPV-18, Month 12: number analyzed (Participants) | 98 | 92 | 98
  Anti-HPV-18, Month 12 | 3546.9 [2829.7 to 4445.8] | 670.3 [510.0 to 880.9] | 1801.4 [1333.0 to 2434.2]
  Anti-HPV-16, Month 18: number analyzed (Participants) | 98 | 90 | 97
  Anti-HPV-16, Month 18 | 7508.8 [5819.8 to 9688.0] | 2070.2 [1494.9 to 2866.9] | 2961.5 [2233.9 to 3926.2]
  Anti-HPV-18, Month 18: number analyzed (Participants) | 97 | 92 | 98
  Anti-HPV-18, Month 18 | 2240.5 [1763.3 to 2846.9] | 294.5 [219.5 to 395.1] | 797.6 [576.3 to 1104.0]
  Anti-HPV-16, Month 24: number analyzed (Participants) | 96 | 87 | 98
  Anti-HPV-16, Month 24 | 4609.1 [3673.5 to 5782.9] | 1193.9 [889.6 to 1602.3] | 1932.0 [1499.4 to 2489.5]
  Anti-HPV-18, Month 24: number analyzed (Participants) | 96 | 87 | 98
  Anti-HPV-18, Month 24 | 1638.6 [1297.9 to 2068.8] | 239.7 [181.2 to 317.1] | 564.6 [418.1 to 762.5]
  Anti-HPV-16, Month 36: number analyzed (Participants) | 98 | 90 | 98
  Anti-HPV-16, Month 36 | 4011.7 [3229.7 to 4983.0] | 1111.4 [849.1 to 1454.6] | 1517.2 [1174.7 to 1959.4]
  Anti-HPV-18, Month 36: number analyzed (Participants) | 97 | 92 | 98
  Anti-HPV-18, Month 36 | 1513.7 [1197.5 to 1913.2] | 185.8 [142.2 to 242.7] | 468.6 [346.3 to 634.0]

11. Secondary Outcome: T-cell-mediated Immune Responses in the Sub-cohort for Cell-Mediated Immunity (CMI)
Description: Among immune markers expressed were Interleukin-2 (IL-2), Interferon-gamma (IFN-γ), Tumour necrosis factor-alpha (TNF-α) and CD40-ligand (CD40-L). The assay was performed on a sub-cohort of approximately 100 subjects per study group.
Time Frame: At Day 0 and Months 7, 12, 24 and 36
Population: The analysis was based on the Month 36 ATP cohort for immunogenicity, which included a sub-cohort of approximately 100 subjects per study group, who returned for blood sampling at Month 36 and for whom data concerning immunogenicity outcome measures were available at the specified time point.
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 67 | 60 | 74
T-cells/million cells
  CD4+ All doubles, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD4+ All doubles, Anti-HPV-16, Day 0 | 10 [1 to 78] | 22 [1 to 90] | 33 [1 to 80]
  CD4+ All doubles, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD4+ All doubles, Anti-HPV-18, Day 0 | 28 [1 to 83] | 47.5 [1 to 102] | 26 [1 to 92]
  CD4+ All doubles, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD4+ All doubles, Anti-HPV-16, Month 7 | 1662 [644 to 3221] | 872 [479 to 1275] | 1121 [694 to 1890]
  CD4+ All doubles, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD4+ All doubles, Anti-HPV-18, Month 7 | 897 [496 to 2497] | 427 [259 to 744] | 640 [355 to 1304]
  CD4+ All doubles, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD4+ All doubles, Anti-HPV-16, Month 12 | 916 [641 to 2340] | 585.5 [316 to 1250] | 819.5 [554 to 1623]
  CD4+ All doubles, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD4+ All doubles, Anti-HPV-18, Month 12 | 789 [384 to 1492] | 327 [184 to 658] | 446 [205 to 824]
  CD4+ All doubles, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD4+ All doubles, Anti-HPV-16, Month 24 | 1068.5 [495 to 2410] | 750.5 [366.5 to 1142.5] | 968.5 [588 to 1830]
  CD4+ All doubles, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD4+ All doubles, Anti-HPV-18, Month 24 | 645 [311 to 1406] | 352 [196.5 to 503] | 578 [267 to 972]
  CD4+ All doubles, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD4+ All doubles, Anti-HPV-16, Month 36 | 1012 [427 to 2373] | 685 [385 to 1321] | 842.5 [437.5 to 1624]
  CD4+ All doubles, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD4+ All doubles, Anti-HPV-18, Month 36 | 682 [313 to 1425] | 350 [196 to 665] | 516 [270 to 1029]
  CD4-d-CD40L, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD4-d-CD40L, Anti-HPV-16, Day 0 | 1 [1 to 73] | 14 [1 to 72] | 30 [1 to 73]
  CD4-d-CD40L, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD4-d-CD40L, Anti-HPV-18, Day 0 | 14 [1 to 83] | 39.5 [1 to 102] | 27.5 [1 to 70]
  CD4-d-CD40L, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD4-d-CD40L, Anti-HPV-16, Month 7 | 1515 [638 to 3098] | 779 [456 to 1211] | 1025.5 [670 to 1848]
  CD4-d-CD40L, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD4-d-CD40L, Anti-HPV-18, Month 7 | 866 [496 to 2483] | 386.5 [237 to 708] | 574 [328 to 1224]
  CD4-d-CD40L, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD4-d-CD40L, Anti-HPV-16, Month 12 | 889 [591 to 2236] | 524 [280 to 1135] | 761.5 [484 to 1425]
  CD4-d-CD40L, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD4-d-CD40L, Anti-HPV-18, Month 12 | 688 [344 to 1435] | 317 [147 to 633] | 383.5 [214 to 729]
  CD4-d-CD40L, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD4-d-CD40L, Anti-HPV-16, Month 24 | 1045.5 [518 to 2269] | 736 [348 to 1101.5] | 937 [588 to 1801]
  CD4-d-CD40L, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD4-d-CD40L, Anti-HPV-18, Month 24 | 639 [310 to 1374] | 332 [204 to 510.5] | 564 [289 to 940]
  CD4-d-CD40L, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD4-d-CD40L, Anti-HPV-16, Month 36 | 957 [465 to 2303] | 685 [349 to 1321] | 778.5 [416.5 to 1560.5]
  CD4-d-CD40L, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD4-d-CD40L, Anti-HPV-18, Month 36 | 671 [290 to 1435] | 337 [204 to 648] | 499 [264 to 1020]
  CD4-d- IFNγ, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD4-d- IFNγ, Anti-HPV-16, Day 0 | 12 [1 to 30] | 19 [1 to 42] | 1 [1 to 28]
  CD4-d- IFNγ, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD4-d- IFNγ, Anti-HPV-18, Day 0 | 14 [1 to 33] | 13.5 [1 to 36] | 3.5 [1 to 30]
  CD4-d- IFNγ, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD4-d- IFNγ, Anti-HPV-16, Month 7 | 365 [161 to 881] | 320 [157 to 533] | 422.5 [206 to 708]
  CD4-d- IFNγ, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD4-d- IFNγ, Anti-HPV-18, Month 7 | 242 [111 to 712] | 133.5 [83 to 240] | 181 [78 to 409]
  CD4-d- IFNγ, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD4-d- IFNγ, Anti-HPV-16, Month 12 | 326 [110 to 644] | 235 [108 to 501] | 356 [135 to 734]
  CD4-d- IFNγ, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD4-d- IFNγ, Anti-HPV-18, Month 12 | 175 [87 to 444] | 112 [55 to 240] | 164 [57 to 315]
  CD4-d- IFNγ, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD4-d- IFNγ, Anti-HPV-16, Month 24 | 300.5 [119 to 781] | 317.5 [146.5 to 514] | 421 [157 to 767]
  CD4-d- IFNγ, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD4-d- IFNγ, Anti-HPV-18, Month 24 | 171 [68 to 462] | 112 [49.5 to 229.5] | 220 [65 to 348]
  CD4-d-IFNγ, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD4-d-IFNγ, Anti-HPV-16, Month 36 | 253.5 [81 to 667] | 301 [134 to 571] | 270.5 [129 to 666.5]
  CD4-d-IFNγ, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD4-d-IFNγ, Anti-HPV-18, Month 36 | 193 [51 to 376] | 109 [27 to 230] | 155 [45 to 314]
  CD4-d-IL-2, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD4-d-IL-2, Anti-HPV-16, Day 0 | 14 [1 to 52] | 25 [1 to 72] | 33 [1 to 56]
  CD4-d-IL-2, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD4-d-IL-2, Anti-HPV-18, Day 0 | 1 [1 to 49] | 36.5 [1 to 76] | 22 [1 to 60]
  CD4-d-IL-2, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD4-d-IL-2, Anti-HPV-16, Month 7 | 1357 [537 to 2660] | 712.5 [378 to 1037] | 866 [561 to 1420]
  CD4-d-IL-2, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD4-d-IL-2, Anti-HPV-18, Month 7 | 737 [420 to 2185] | 304 [206 to 573] | 486 [281 to 959]
  CD4-d-IL-2, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD4-d-IL-2, Anti-HPV-16, Month 12 | 832 [493 to 2050] | 479 [283 to 946] | 674.5 [450 to 1316]
  CD4-d-IL-2, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD4-d-IL-2, Anti-HPV-18, Month 12 | 620 [304 to 1157] | 259 [144 to 547] | 354 [155 to 622]
  CD4-d-IL-2, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD4-d-IL-2, Anti-HPV-16, Month 24 | 855 [390 to 1711] | 579.5 [270.5 to 934.5] | 700 [479 to 1459]
  CD4-d-IL-2, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD4-d-IL-2, Anti-HPV-18, Month 24 | 494 [252 to 994] | 240 [125.5 to 387.5] | 426 [216 to 695]
  CD4-d-IL-2, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD4-d-IL-2, Anti-HPV-16, Month 36 | 784 [331 to 1673] | 517 [295 to 1014] | 680 [308 to 1245.5]
  CD4-d-IL-2, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD4-d-IL-2, Anti-HPV-18, Month 36 | 507 [213 to 1069] | 274 [137 to 467] | 341 [168 to 798]
  CD4-d-TNFα, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD4-d-TNFα, Anti-HPV-16, Day 0 | 6 [1 to 50] | 33 [1 to 82] | 16 [1 to 69]
  CD4-d-TNFα, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD4-d-TNFα, Anti-HPV-18, Day 0 | 27 [1 to 75] | 22.5 [1 to 82] | 23 [1 to 60]
  CD4-d-TNFα, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD4-d-TNFα, Anti-HPV-16, Month 7 | 1111 [430 to 2386] | 625 [292 to 899] | 796 [458 to 1448]
  CD4-d-TNFα, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD4-d-TNFα, Anti-HPV-18, Month 7 | 647 [336 to 1415] | 283.5 [168 to 594] | 457 [266 to 978]
  CD4-d-TNFα, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD4-d-TNFα, Anti-HPV-16, Month 12 | 790 [488 to 1924] | 482 [210 to 932] | 716 [457 to 1445]
  CD4-d-TNFα, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD4-d-TNFα, Anti-HPV-18, Month 12 | 674 [288 to 1272] | 266 [133 to 588] | 384.5 [175 to 714]
  CD4-d-TNFα, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD4-d-TNFα, Anti-HPV-16, Month 24 | 795.5 [343 to 1668] | 563.5 [241.5 to 895] | 760.5 [443 to 1494]
  CD4-d-TNFα, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD4-d-TNFα, Anti-HPV-18, Month 24 | 510 [183 to 1164] | 239 [127.5 to 440.5] | 522 [228 to 710]
  CD4-d-TNFα, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD4-d-TNFα, Anti-HPV-16, Month 36 | 786.5 [343 to 1930] | 547 [282 to 1005] | 724.5 [368 to 1338]
  CD4-d-TNFα, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD4-d-TNFα, Anti-HPV-18, Month 36 | 588 [250 to 1138] | 301 [120 to 453] | 479 [200 to 808]
  CD8-All Doubles, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD8-All Doubles, Anti-HPV-16, Day 0 | 1 [1 to 14] | 4 [1 to 49] | 1 [1 to 25]
  CD8-All Doubles, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD8-All Doubles, Anti-HPV-18, Day 0 | 1 [1 to 16] | 1 [1 to 29] | 1 [1 to 22]
  CD8-All Doubles, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD8-All Doubles, Anti-HPV-16, Month 7 | 1 [1 to 34] | 1 [1 to 41] | 1 [1 to 30]
  CD8-All Doubles, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD8-All Doubles, Anti-HPV-18, Month 7 | 1 [1 to 19] | 1 [1 to 40] | 1 [1 to 40]
  CD8-All Doubles, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD8-All Doubles, Anti-HPV-16, Month 12 | 1 [1 to 31] | 1 [1 to 29] | 1 [1 to 29]
  CD8-All Doubles, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD8-All Doubles, Anti-HPV-18, Month 12 | 1 [1 to 27] | 1 [1 to 27] | 1 [1 to 20]
  CD8-All Doubles, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD8-All Doubles, Anti-HPV-16, Month 24 | 1 [1 to 25] | 1 [1 to 1] | 1 [1 to 1]
  CD8-All Doubles, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD8-All Doubles, Anti-HPV-18, Month 24 | 1 [1 to 32] | 1 [1 to 23] | 1 [1 to 28]
  CD8-All doubles, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD8-All doubles, Anti-HPV-16, Month 36 | 1 [1 to 48] | 1 [1 to 28] | 1 [1 to 38.5]
  CD8-All doubles, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD8-All doubles, Anti-HPV-18, Month 36 | 4 [1 to 40] | 2 [1 to 41] | 1 [1 to 28]
  CD8-d-CD40L, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD8-d-CD40L, Anti-HPV-16, Day 0 | 1 [1 to 1] | 1 [1 to 26] | 1 [1 to 1]
  CD8-d-CD40L, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD8-d-CD40L, Anti-HPV-18, Day 0 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-CD40L, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD8-d-CD40L, Anti-HPV-16, Month 7 | 1 [1 to 1] | 1 [1 to 29] | 1 [1 to 24]
  CD8-d-CD40L, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD8-d-CD40L, Anti-HPV-18, Month 7 | 1 [1 to 1] | 1 [1 to 24] | 1 [1 to 23]
  CD8-d-CD40L, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD8-d-CD40L, Anti-HPV-16, Month 12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 3]
  CD8-d-CD40L, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD8-d-CD40L, Anti-HPV-18, Month 12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-CD40L, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD8-d-CD40L, Anti-HPV-16, Month 24 | 1 [1 to 16] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-CD40L, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD8-d-CD40L, Anti-HPV-18, Month 24 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 18]
  CD8-d-CD40L, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD8-d-CD40L, Anti-HPV-16, Month 36 | 1 [1 to 31] | 1 [1 to 24] | 1 [1 to 29]
  CD8-d-CD40L, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD8-d-CD40L, Anti-HPV-18, Month 36 | 1 [1 to 6] | 1 [1 to 27] | 1 [1 to 28]
  CD8-d-IFNγ, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD8-d-IFNγ, Anti-HPV-16, Day 0 | 1 [1 to 1] | 1 [1 to 39] | 1 [1 to 26]
  CD8-d-IFNγ, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD8-d-IFNγ, Anti-HPV-18, Day 0 | 1 [1 to 2] | 1 [1 to 23] | 1 [1 to 18]
  CD8-d-IFNγ, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD8-d-IFNγ, Anti-HPV-16, Month 7 | 1 [1 to 32] | 1 [1 to 40] | 1 [1 to 30]
  CD8-d-IFNγ, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD8-d-IFNγ, Anti-HPV-18, Month 7 | 1 [1 to 1] | 1 [1 to 28] | 1 [1 to 28]
  CD8-d-IFNγ, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD8-d-IFNγ, Anti-HPV-16, Month 12 | 1 [1 to 28] | 1 [1 to 26] | 1 [1 to 27]
  CD8-d-IFNγ, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD8-d-IFNγ, Anti-HPV-18, Month 12 | 1 [1 to 22] | 1 [1 to 26] | 1 [1 to 10]
  CD8-d-IFNγ, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD8-d-IFNγ, Anti-HPV-16, Month 24 | 1 [1 to 16] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IFNγ, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD8-d-IFNγ, Anti-HPV-18, Month 24 | 1 [1 to 18] | 1 [1 to 23] | 1 [1 to 1]
  CD8-d-IFNγ, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD8-d-IFNγ, Anti-HPV-16, Month 36 | 1 [1 to 47] | 1 [1 to 25] | 1 [1 to 33]
  CD8-d-IFNγ, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD8-d-IFNγ, Anti-HPV-18, Month 36 | 1 [1 to 31] | 2 [1 to 40] | 1 [1 to 25]
  CD8-d-IL-2, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD8-d-IL-2, Anti-HPV-16, Day 0 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IL-2, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD8-d-IL-2, Anti-HPV-18, Day 0 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IL-2, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD8-d-IL-2, Anti-HPV-16, Month 7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IL-2, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD8-d-IL-2, Anti-HPV-18, Month 7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IL-2, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD8-d-IL-2, Anti-HPV-16, Month 12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IL-2, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD8-d-IL-2, Anti-HPV-18, Month 12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IL-2, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD8-d-IL-2, Anti-HPV-16, Month 24 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IL-2, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD8-d-IL-2, Anti-HPV-18, Month 24 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IL-2, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD8-d-IL-2, Anti-HPV-16, Month 36 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-IL-2, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD8-d-IL-2, Anti-HPV-18, Month 36 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-TNFα, Anti-HPV-16, Day 0: number analyzed (Participants) | 53 | 42 | 53
  CD8-d-TNFα, Anti-HPV-16, Day 0 | 1 [1 to 1] | 1 [1 to 36] | 1 [1 to 16]
  CD8-d-TNFα, Anti-HPV-18, Day 0: number analyzed (Participants) | 53 | 42 | 54
  CD8-d-TNFα, Anti-HPV-18, Day 0 | 1 [1 to 27] | 1 [1 to 29] | 1 [1 to 26]
  CD8-d-TNFα, Anti-HPV-16, Month 7: number analyzed (Participants) | 63 | 58 | 62
  CD8-d-TNFα, Anti-HPV-16, Month 7 | 1 [1 to 28] | 1 [1 to 26] | 1 [1 to 18]
  CD8-d-TNFα, Anti-HPV-18, Month 7: number analyzed (Participants) | 63 | 58 | 63
  CD8-d-TNFα, Anti-HPV-18, Month 7 | 1 [1 to 1] | 1 [1 to 2] | 1 [1 to 24]
  CD8-d-TNFα, Anti-HPV-16, Month 12: number analyzed (Participants) | 67 | 58 | 66
  CD8-d-TNFα, Anti-HPV-16, Month 12 | 1 [1 to 1] | 1 [1 to 25] | 1 [1 to 28]
  CD8-d-TNFα, Anti-HPV-18, Month 12: number analyzed (Participants) | 67 | 59 | 66
  CD8-d-TNFα, Anti-HPV-18, Month 12 | 1 [1 to 8] | 1 [1 to 21] | 1 [1 to 24]
  CD8-d-TNFα, Anti-HPV-16, Month 24: number analyzed (Participants) | 66 | 60 | 74
  CD8-d-TNFα, Anti-HPV-16, Month 24 | 1 [1 to 20] | 1 [1 to 1] | 1 [1 to 1]
  CD8-d-TNFα, Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 60 | 73
  CD8-d-TNFα, Anti-HPV-18, Month 24 | 1 [1 to 28] | 1 [1 to 7] | 1 [1 to 18]
  CD8-d-TNFα, Anti-HPV-16, Month 36: number analyzed (Participants) | 58 | 55 | 64
  CD8-d-TNFα, Anti-HPV-16, Month 36 | 1 [1 to 24] | 1 [1 to 1] | 1 [1 to 26]
  CD8-d-TNFα, Anti-HPV-18, Month 36: number analyzed (Participants) | 57 | 55 | 63
  CD8-d-TNFα, Anti-HPV-18, Month 36 | 1 [1 to 31] | 1 [1 to 21] | 1 [1 to 12]

12. Secondary Outcome: B-cell-mediated Immune Responses in the Sub-cohort for CMI
Description: The frequency of B-cell Elispot response to HPV-16/18 by overall status was presented. The assay was performed on a sub-cohort of approximately 100 subjects per study group.
Time Frame: At Day 0 and Months 7, 12, 24 and 36
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: B-cells/million cells
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 71 | 65 | 76
B-cells/million cells
  HPV-16, Day 0: number analyzed (Participants) | 69 | 55 | 70
  HPV-16, Day 0 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HPV-18, Day 0: number analyzed (Participants) | 69 | 55 | 70
  HPV-18, Day 0 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HPV-16, Month 7 | 1733 [577 to 3733] | 1254 [495 to 2173] | 733 [106.5 to 1966.5]
  HPV-18, Month 7 | 558 [106 to 1847] | 155 [1 to 379] | 111 [1 to 343.5]
  HPV-16, Month 12: number analyzed (Participants) | 51 | 51 | 53
  HPV-16, Month 12 | 408 [90 to 1186] | 278 [66 to 794] | 289 [66 to 982]
  HPV-18, Month 12: number analyzed (Participants) | 51 | 51 | 53
  HPV-18, Month 12 | 249 [73 to 658] | 69 [1 to 184] | 69 [1 to 250]
  HPV-16, Month 24: number analyzed (Participants) | 54 | 46 | 63
  HPV-16, Month 24 | 270 [49 to 724] | 218.5 [28 to 651] | 249 [37 to 601]
  HPV-18, Month 24: number analyzed (Participants) | 54 | 46 | 63
  HPV-18, Month 24 | 128.5 [35 to 402] | 57.5 [1 to 203] | 111 [1 to 317]
  HPV-16, Month 36: number analyzed (Participants) | 59 | 54 | 53
  HPV-16, Month 36 | 353 [91 to 927] | 382.5 [166 to 614] | 246 [21 to 565]
  HPV-18, Month 36: number analyzed (Participants) | 59 | 54 | 53
  HPV-18, Month 36 | 116 [1 to 329] | 25 [1 to 228] | 63 [1 to 150]

13. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimetres (mm) of injection site.
Time Frame: During the 7-day period (from the day of vaccination up to 6 subsequent days) following vaccination after each dose and across doses
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered and who had their symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 359 | 357 | 356
Participants
  Any Pain - Dose 1 | 311 | 235 | 231
  Any Pain - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Pain - Dose 2 | 193 | 183 | 215
  Any Pain - Dose 3: number analyzed (Participants) | 356 | 348 | 350
  Any Pain - Dose 3 | 280 | 194 | 222
  Any Pain - Across doses | 329 | 276 | 295
  Grade 3 Pain - Dose 1 | 22 | 4 | 6
  Grade 3 Pain - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Pain - Dose 2 | 8 | 8 | 8
  Grade 3 Pain - Dose 3: number analyzed (Participants) | 356 | 348 | 350
  Grade 3 Pain - Dose 3 | 23 | 11 | 10
  Grade 3 Pain - Across doses | 42 | 17 | 18
  Any Redness - Dose 1 | 137 | 84 | 87
  Any Redness - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Redness - Dose 2 | 100 | 84 | 99
  Any Redness - Dose 3: number analyzed (Participants) | 356 | 348 | 350
  Any Redness - Dose 3 | 133 | 92 | 102
  Any Redness - Across doses | 191 | 134 | 157
  Grade 3 Redness - Dose 1 | 0 | 0 | 1
  Grade 3 Redness - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Redness - Dose 2 | 0 | 0 | 0
  Grade 3 Redness - Dose 3: number analyzed (Participants) | 356 | 348 | 350
  Grade 3 Redness - Dose 3 | 0 | 0 | 1
  Grade 3 Redness - Across doses | 0 | 0 | 2
  Any Swelling - Dose 1 | 112 | 44 | 39
  Any Swelling - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Swelling - Dose 2 | 63 | 35 | 76
  Any Swelling - Dose 3: number analyzed (Participants) | 356 | 348 | 350
  Any Swelling - Dose 3 | 113 | 67 | 85
  Any Swelling - Across doses | 163 | 98 | 118
  Grade 3 Swelling - Dose 1 | 3 | 0 | 0
  Grade 3 Swelling - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Swelling - Dose 2 | 0 | 0 | 0
  Grade 3 Swelling - Dose 3: number analyzed (Participants) | 356 | 348 | 350
  Grade 3 Swelling - Dose 3 | 2 | 0 | 2
  Grade 3 Swelling - Across doses | 5 | 0 | 2

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, rash, temperature [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)] and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever above (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 359 | 357 | 356
Participants
  Any Arthralgia - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Any Arthralgia - Dose 1 | 44 | 50 | 39
  Any Arthralgia - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Arthralgia - Dose 2 | 23 | 30 | 34
  Any Arthralgia - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Any Arthralgia - Dose 3 | 31 | 38 | 35
  Any Arthralgia - Across doses | 68 | 81 | 67
  Grade 3 Arthralgia - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Grade 3 Arthralgia - Dose 1 | 5 | 1 | 1
  Grade 3 Arthralgia - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Arthralgia - Dose 2 | 1 | 2 | 1
  Grade 3 Arthralgia - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Grade 3 Arthralgia - Dose 3 | 2 | 3 | 1
  Grade 3 Arthralgia - Across doses | 6 | 4 | 1
  Related Arthralgia - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Related Arthralgia - Dose 1 | 29 | 32 | 28
  Related Arthralgia - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Related Arthralgia - Dose 2 | 17 | 17 | 18
  Related Arthralgia - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Related Arthralgia - Dose 3 | 20 | 27 | 27
  Related Arthralgia - Across doses | 51 | 55 | 51
  Any Fatigue - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Any Fatigue - Dose 1 | 163 | 157 | 168
  Any Fatigue - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Fatigue - Dose 2 | 103 | 104 | 119
  Any Fatigue - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Any Fatigue - Dose 3 | 108 | 97 | 103
  Any Fatigue - Across doses | 192 | 199 | 193
  Grade 3 Fatigue - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Grade 3 Fatigue - Dose 1 | 7 | 10 | 5
  Grade 3 Fatigue - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Fatigue - Dose 2 | 12 | 3 | 2
  Grade 3 Fatigue - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Grade 3 Fatigue - Dose 3 | 7 | 3 | 3
  Grade 3 Fatigue - Across doses | 18 | 15 | 7
  Related Fatigue - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Related Fatigue - Dose 1 | 103 | 102 | 98
  Related Fatigue - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Related Fatigue - Dose 2 | 68 | 66 | 67
  Related Fatigue - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Related Fatigue - Dose 3 | 70 | 67 | 67
  Related Fatigue - Across doses | 152 | 151 | 143
  Any Gastrointestinal - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Any Gastrointestinal - Dose 1 | 34 | 52 | 44
  Any Gastrointestinal - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Gastrointestinal - Dose 2 | 19 | 22 | 23
  Any Gastrointestinal - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Any Gastrointestinal - Dose 3 | 16 | 29 | 24
  Any Gastrointestinal - Across doses | 55 | 74 | 70
  Grade 3 Gastrointestinal - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Grade 3 Gastrointestinal - Dose 1 | 3 | 2 | 2
  Grade 3 Gastrointestinal - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Gastrointestinal - Dose 2 | 2 | 1 | 0
  Grade 3 Gastrointestinal - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Grade 3 Gastrointestinal - Dose 3 | 1 | 4 | 2
  Grade 3 Gastrointestinal - Across doses | 5 | 6 | 3
  Related Gastrointestinal - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Related Gastrointestinal - Dose 1 | 21 | 26 | 22
  Related Gastrointestinal - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Related Gastrointestinal - Dose 2 | 8 | 17 | 6
  Related Gastrointestinal - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Related Gastrointestinal - Dose 3 | 10 | 20 | 17
  Related Gastrointestinal - Across doses | 32 | 49 | 40
  Any Headache - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Any Headache - Dose 1 | 102 | 87 | 90
  Any Headache - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Headache - Dose 2 | 62 | 64 | 73
  Any Headache - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Any Headache - Dose 3 | 63 | 54 | 65
  Any Headache - Across doses | 147 | 133 | 151
  Grade 3 Headache - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Grade 3 Headache - Dose 1 | 7 | 6 | 1
  Grade 3 Headache - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Headache - Dose 2 | 6 | 2 | 4
  Grade 3 Headache - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Grade 3 Headache - Dose 3 | 7 | 1 | 1
  Grade 3 Headache - Across doses | 17 | 7 | 4
  Related Headache - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Related Headache - Dose 1 | 61 | 51 | 48
  Related Headache - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Related Headache - Dose 2 | 39 | 37 | 41
  Related Headache - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Related Headache - Dose 3 | 45 | 33 | 42
  Related Headache - Across doses | 107 | 88 | 100
  Any Myalgia - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Any Myalgia - Dose 1 | 131 | 101 | 101
  Any Myalgia - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Myalgia - Dose 2 | 59 | 60 | 80
  Any Myalgia - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Any Myalgia - Dose 3 | 77 | 68 | 72
  Any Myalgia - Across doses | 166 | 143 | 136
  Grade 3 Myalgia - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Grade 3 Myalgia - Dose 1 | 5 | 3 | 2
  Grade 3 Myalgia - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Myalgia - Dose 2 | 2 | 3 | 2
  Grade 3 Myalgia - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Grade 3 Myalgia - Dose 3 | 3 | 4 | 5
  Grade 3 Myalgia - Across doses | 8 | 8 | 6
  Related Myalgia - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Related Myalgia - Dose 1 | 91 | 70 | 67
  Related Myalgia - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Related Myalgia - Dose 2 | 36 | 40 | 51
  Related Myalgia - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Related Myalgia - Dose 3 | 50 | 49 | 46
  Related Myalgia - Across doses | 128 | 111 | 100
  Any Rash - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Any Rash - Dose 1 | 14 | 7 | 10
  Any Rash - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Rash - Dose 2 | 10 | 5 | 8
  Any Rash - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Any Rash - Dose 3 | 7 | 5 | 4
  Any Rash - Across doses | 25 | 16 | 18
  Grade 3 Rash - Dose 1 | 0 | 0 | 0
  Grade 3 Rash - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Rash - Dose 2 | 0 | 0 | 0
  Grade 3 Rash - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Grade 3 Rash - Dose 3 | 0 | 0 | 0
  Grade 3 Rash - Across doses | 0 | 0 | 0
  Related Rash - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Related Rash - Dose 1 | 6 | 5 | 6
  Related Rash - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Related Rash - Dose 2 | 6 | 3 | 4
  Related Rash - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Related Rash - Dose 3 | 6 | 3 | 3
  Related Rash - Across doses | 16 | 10 | 12
  Any Temperature ( ≥ 37.5°C) - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Any Temperature ( ≥ 37.5°C) - Dose 1 | 19 | 23 | 18
  Any Temperature ( ≥ 37.5°C) - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Temperature ( ≥ 37.5°C) - Dose 2 | 13 | 21 | 19
  Any Temperature ( ≥ 37.5°C) - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Any Temperature ( ≥ 37.5°C) - Dose 3 | 32 | 22 | 22
  Any Temperature ( ≥ 37.5°C) - Across doses | 53 | 59 | 47
  Grade 3 Temperature ( > 39.0°C) - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Grade 3 Temperature ( > 39.0°C) - Dose 1 | 2 | 2 | 2
  Grade 3 Temperature ( > 39.0°C) - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Temperature ( > 39.0°C) - Dose 2 | 0 | 0 | 2
  Grade 3 Temperature ( > 39.0°C) - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Grade 3 Temperature ( > 39.0°C) - Dose 3 | 6 | 0 | 0
  Grade 3 Temperature ( > 39.0°C) - Across doses | 7 | 2 | 4
  Related Temperature - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Related Temperature - Dose 1 | 13 | 11 | 7
  Related Temperature - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Related Temperature - Dose 2 | 8 | 9 | 11
  Related Temperature - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Related Temperature - Dose 3 | 19 | 12 | 15
  Related Temperature - Across doses | 35 | 31 | 30
  Any Urticaria - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Any Urticaria - Dose 1 | 15 | 7 | 12
  Any Urticaria - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Any Urticaria - Dose 2 | 8 | 5 | 12
  Any Urticaria - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Any Urticaria - Dose 3 | 11 | 4 | 9
  Any Urticaria - Across doses | 28 | 13 | 25
  Grade 3 Urticaria - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Grade 3 Urticaria - Dose 1 | 2 | 0 | 0
  Grade 3 Urticaria - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Grade 3 Urticaria - Dose 2 | 0 | 1 | 0
  Grade 3 Urticaria - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Grade 3 Urticaria - Dose 3 | 2 | 0 | 0
  Grade 3 Urticaria - Across doses | 4 | 1 | 0
  Related Urticaria - Dose 1: number analyzed (Participants) | 359 | 357 | 355
  Related Urticaria - Dose 1 | 7 | 6 | 7
  Related Urticaria - Dose 2: number analyzed (Participants) | 357 | 353 | 354
  Related Urticaria - Dose 2 | 5 | 4 | 4
  Related Urticaria - Dose 3: number analyzed (Participants) | 354 | 347 | 351
  Related Urticaria - Dose 3 | 6 | 4 | 2
  Related Urticaria - Across doses | 15 | 11 | 9

15. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (from the day of vaccination up to 29 subsequent days) post-vaccination period
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 359 | 358 | 358
Participants
  Subjects with any AE(s) | 91 | 96 | 101
  Subjects with any Grade 3 AE(s) | 18 | 8 | 20
  Subjects with any Related AE(s) | 8 | 14 | 15

16. Secondary Outcome: Number of Subjects With Potentially Immune Mediated Diseases (pIMDs)
Description: pIMDs were defined as a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Day 0 up to Month 12
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 359 | 358 | 358
Participants | 3 | 3 | 0

17. Secondary Outcome: Number of Subjects With Medically Significant Conditions (MSCs)
Description: MSCs were defined as AEs prompting emergency room (ER) or physician visits that were not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or SAEs not related to common diseases. Common diseases include: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From Day 0 up to Month 36 (throughout the study period)
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 359 | 358 | 358
Participants | 77 | 79 | 63

18. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: From Day 0 up to Month 36 (throughout the study period)
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 359 | 358 | 358
Participants | 21 | 11 | 14

19. Secondary Outcome: Number of Subjects With SAEs Related to the Investigational Product, to Study Participation, to GSK Concomitant Products or Any Fatal SAE
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Related = an event assessed by the investigator as causally related to the investigational product, to study participation or to GSK concomitant products.
Time Frame: From Day 0 up to Month 36 (throughout the study period)
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 359 | 358 | 358
Participants
  Related SAE(s) | 0 | 0 | 0
  Fatal SAE(s) | 0 | 0 | 1

20. Secondary Outcome: Number of Subjects Reporting Pregnancies and Outcomes of Reported Pregnancies
Description: Outcomes of pregnancies were Live infant NO apparent congenital anomaly (ACA), Live infant congenital anomaly (CA), Elective termination NO ACA, Elective termination CA, Ectopic pregnancy, Spontaneous abortion NO ACA, Stillbirth NO ACA, Stillbirth CA, Lost to follow up and Pregnancy ongoing.
Time Frame: From Day 0 up to Month 36 (throughout the study period)
Population: The analysis was based on the TVC, which included all subjects with the study vaccine administered and who reported any pregnancies and outcomes of reported pregnancies.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 0 | 0 | 1
Participants
  Live infant NO ACA: number analyzed (Participants) | 0 | 0 | 0
  Live infant NO ACA | 0 | 0 | 0
  Live infant CA: number analyzed (Participants) | 0 | 0 | 0
  Live infant CA | 0 | 0 | 0
  Elective termination NO ACA | 0 | 0 | 1
  Elective termination CA: number analyzed (Participants) | 0 | 0 | 0
  Elective termination CA | 0 | 0 | 0
  Ectopic pregnancy: number analyzed (Participants) | 0 | 0 | 0
  Ectopic pregnancy | 0 | 0 | 0
  Spontaneous abortion NO ACA: number analyzed (Participants) | 0 | 0 | 0
  Spontaneous abortion NO ACA | 0 | 0 | 0
  Stillbirth NO ACA: number analyzed (Participants) | 0 | 0 | 0
  Stillbirth NO ACA | 0 | 0 | 0
  Stillbirth CA: number analyzed (Participants) | 0 | 0 | 0
  Stillbirth CA | 0 | 0 | 0
  Lost to follow up: number analyzed (Participants) | 0 | 0 | 0
  Lost to follow up | 0 | 0 | 0
  Pregnancy ongoing: number analyzed (Participants) | 0 | 0 | 0
  Pregnancy ongoing | 0 | 0 | 0
  Missing: number analyzed (Participants) | 0 | 0 | 0
  Missing | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects Using a Concomitant Medication Throughout the Study Period
Description: The number of subjects who have used any concomitant medication, as well as any antipyretic, any prophylactic antipyretic and any antibiotic.
Time Frame: From Day 0 up to Month 36 (throughout the study period) following vaccination after each dose and across doses
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 359 | 358 | 358
Participants
  Any, Dose 1 | 85 | 87 | 93
  Any antipyretic, Dose 1 | 51 | 53 | 47
  Prophylactic antipyretic, Dose 1 | 4 | 0 | 0
  Any antibiotic, Dose 1 | 15 | 13 | 23
  Prophylactic antibiotic, Dose 1 | 0 | 0 | 0
  Any, Dose 2: number analyzed (Participants) | 358 | 356 | 356
  Any, Dose 2 | 52 | 55 | 47
  Any antipyretic, Dose 2: number analyzed (Participants) | 358 | 356 | 356
  Any antipyretic, Dose 2 | 32 | 26 | 29
  Prophylactic antipyretic, Dose 2: number analyzed (Participants) | 358 | 356 | 356
  Prophylactic antipyretic, Dose 2 | 0 | 1 | 2
  Any antibiotic, Dose 2: number analyzed (Participants) | 358 | 356 | 356
  Any antibiotic, Dose 2 | 8 | 13 | 12
  Prophylactic antibiotic, Dose 2: number analyzed (Participants) | 358 | 356 | 356
  Prophylactic antibiotic, Dose 2 | 0 | 0 | 0
  Any, Dose 3: number analyzed (Participants) | 357 | 352 | 354
  Any, Dose 3 | 90 | 83 | 81
  Any antipyretic, Dose 3: number analyzed (Participants) | 357 | 352 | 354
  Any antipyretic, Dose 3 | 48 | 45 | 38
  Prophylactic antipyretic, Dose 3: number analyzed (Participants) | 357 | 352 | 354
  Prophylactic antipyretic, Dose 3 | 3 | 1 | 0
  Any antibiotic, Dose 3: number analyzed (Participants) | 357 | 352 | 354
  Any antibiotic, Dose 3 | 28 | 21 | 24
  Prophylactic antibiotic, Dose 3: number analyzed (Participants) | 357 | 352 | 354
  Prophylactic antibiotic, Dose 3 | 0 | 0 | 0
  Any, Across doses | 171 | 157 | 161
  Any antipyretic, Across doses | 110 | 102 | 95
  Prophylactic antipyretic, Across doses | 5 | 2 | 2
  Any antibiotic, Across doses | 48 | 42 | 50
  Prophylactic antibiotic, Across doses | 0 | 0 | 0

22. Secondary Outcome: Number of Subjects Completing the Vaccination Schedule
Description: The number of subjects who have completed the three-dose vaccination schedule in all groups.
Time Frame: From Day 0 up to Month 36 (throughout the study period)
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
Number analyzed (Participants) | 359 | 358 | 358
Participants | 351 | 339 | 346

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day period after vaccination. Unsolicited AEs: during the 30-day period after vaccination. SAEs: throughout the study period (from Day 0 up to Month 36).
Arm/Group | Cervarix 2 Dose Group | Gardasil 2 Dose Group | Gardasil 3 Dose Group
All-Cause Mortality (participants affected / at risk) | 0/359 | 0/358 | 1/358
Serious Adverse Events (participants affected / at risk) | 21/359 | 11/358 | 14/358
Other Adverse Events (participants affected / at risk) | 343/359 | 321/358 | 324/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix 2 Dose Group (N=359) | Gardasil 2 Dose Group (N=358) | Gardasil 3 Dose Group (N=358)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulval ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix 2 Dose Group (N=359) | Gardasil 2 Dose Group (N=358) | Gardasil 3 Dose Group (N=358)
Arthralgia (Musculoskeletal and connective tissue disorders) | 68 (98) | 82 (119) | 67 (108)
Erythema (Skin and subcutaneous tissue disorders) | 191 (370) | 135 (261) | 157 (288)
Fatigue (General disorders) | 192 (374) | 199 (359) | 193 (390)
Gastrointestinal disorder (Gastrointestinal disorders) | 55 (69) | 74 (103) | 70 (91)
Headache (Nervous system disorders) | 149 (241) | 134 (213) | 152 (232)
Myalgia (Musculoskeletal and connective tissue disorders) | 166 (267) | 144 (230) | 136 (254)
Nasopharyngitis (Infections and infestations) | 8 (10) | 11 (12) | 20 (22)
Pain (General disorders) | 329 (784) | 277 (613) | 295 (669)
Pyrexia (General disorders) | 59 (70) | 64 (71) | 53 (65)
Rash (Skin and subcutaneous tissue disorders) | 26 (32) | 16 (17) | 18 (23)
Swelling (General disorders) | 163 (288) | 98 (146) | 118 (200)
Upper respiratory tract infection (Infections and infestations) | 27 (31) | 29 (33) | 31 (34)
Urticaria (Skin and subcutaneous tissue disorders) | 28 (36) | 13 (16) | 25 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.